CLINICAL TRIAL: NCT03289013
Title: A Pilot Evaluation Exploring New Adhesive Materials and Their Ability to Handle Moisture From Abdominal and Peristomal Skin
Brief Title: Assessement of the Peal Force Needed to Peel New Adhesives From the Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CP267_02
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Ileostomy - Stoma
MeSH Terms: interventions — cholecystokinin 33 (10-20)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Testing of new adhesive strips (Experimental): Each subject will test six adhesive strips on pre-stripped skin.
  1. Standard adhesive 1
  2. Standard adhesive 2
  3. LT-2
  4. LT-21
  5. LT-25
  6. 33-20
  The six strips are applied on the abdominal skin. The order of the adhesive strips on the skin is randomized. The subjects will change the adhesive strips at home and the adhesion of adhesive strips will be measured at 5 visits.
  Interventions: Other: Standard adhesive 1; Other: Standard adhesive 2; Other: LT-2; Other: LT-21; Other: LT-25; Other: 33-20

INTERVENTIONS:
Other: Standard adhesive 1 — This strip consists of a standard hydrocolloid adhesive found in ostomy devices
Other: Standard adhesive 2 — This strip consists of a standard hydrocolloid adhesive found in ostomy devices
Other: LT-2 — Newly developed adhesive
Other: LT-21 — Newly developed adhesive
Other: LT-25 — Newly developed adhesive
Other: 33-20 — Newly developed adhesive

SUMMARY:
This study investigates the adhesion of new adhesives to the skin.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be at least 18 years of age and have full legal capacity
3. Have intact skin on the area used in the investigation

Exclusion Criteria:

1. Currently receiving or have within the past 2 months received radio- and/or chemotherapy
2. Currently receiving or have within the past months received topical steroid treatment in the abdominal skin area or systemic steroid (tablet/injection) treatment.
3. Are pregnant or breastfeeding
4. Have dermatological problems in the abdominal area (assessed by investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Swelling of the adhesive | 21 days
  1. Swelling of adhesive strips measured by weight (Difference between weight of strip before and after test)

CONTACTS AND LOCATIONS:
Overall Officials: Lene Feldskov, Principal Investigator — Head of preclinical department
Locations (1):
- Coloplast A/S, Humlebæk, Denmark